CLINICAL TRIAL: NCT00006437
Title: Pathophysiology of Chronic Wounds: Collection of Blood From Healthy Volunteers
Brief Title: Pathophysiology of Chronic Wounds
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010026; 01-D-0026
Record Dates: First submitted 2000-11-03; First posted 2000-11-06 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-10

CONDITIONS: Healthy; Skin Ulcer
Keywords: MMP; Proteases; Adhesion; Migration; Extracellular Matrix
MeSH Terms: conditions — Skin Ulcer; Tissue Adhesions

SUMMARY:
This study will compare blood from healthy volunteers and with wound fluid and tissue samples from patients with acute and chronic wounds enrolled in other NIH studies. Chronic wounds, such as venous leg ulcers, pressure sores, ischemic ulcers and diabetic foot ulcers, affect more than 4 million Americans each year and cost about $9 billion to treat. The nature of these wounds is not well understood and treatments are not always successful, for unknown reasons. Blood collected from healthy volunteers will be used to prepare a model for studying various processes involved in wound healing.

Normal healthy volunteers 21 years of age and older who do not smoke and have no medical problems of the heart, bones, muscles, stomach, lungs, blood, or nervous system, do not have problems going to the bathroom, and have no infections may be eligible for this study.

Participants will be interviewed briefly for information on their date of birth, gender, ethnic identity and medical history and will have a brief physical examination, including a check of height and weight, vital signs and heart and lung sounds. About 14 milliliters (2 tablespoons) of blood will be drawn from the arm.

DETAILED DESCRIPTION:
Chronic wounds are "any interruption on the continuity of the body's tissue that requires a prolonged time to heal, does not heal, or recurs" (Wysocki, 1996). Venous leg ulcers, pressure sores, ischemic ulcers, and diabetic foot ulcers are examples of chronic wounds. These kinds of wounds affect over 4 million Americans each year and cost over $9 billion to treat. The pathophysiology of these wounds is not well understood and therapies directed at healing these wounds are not always successful for unknown reasons. To better understand the pathophysiology of these wounds we propose to collect blood by venipuncture from healthy volunteers. Blood will be used to prepare blood and plasma derived serum for use in an in vitro wound healing model and Boyden chamber assays to study cell migration, adhesion, genetic expression, expression of cell surface receptors, and protein expression to construct a profile of various healing processes. This baseline data will be used for studying the effect of acute and chronic wound fluids on cell migration, adhesion, genetic expression, expression of cell surface receptor and protein expression in an in vitro wound model (protocols to be submitted for each patient population).

ELIGIBILITY:
INCLUSION CRITERIA

Healthy volunteers, 21 years of age and older.

Male or female.

EXCLUSION CRITERIA

Volunteers with known neurological, cardiac, endocrine, skeletal, gastrointestinal, immunological, neoplastic, pulmonary, urologic, hematologic, or infectious disease.

Volunteers taking medications to treat a known diagnosed illness.

Smoker.

Children will not be used because chronic wounds are rarely seen in this population.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 999
Dates: Start 2000-10; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Grinnell F, Ho CH, Wysocki A. Degradation of fibronectin and vitronectin in chronic wound fluid: analysis by cell blotting, immunoblotting, and cell adhesion assays. J Invest Dermatol. 1992 Apr;98(4):410-6. doi: 10.1111/1523-1747.ep12499839. PMID 1372338
- [Background] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Background] Wysocki AB. Surgical wound healing. A review for perioperative nurses. AORN J. 1989 Feb;49(2):502, 504-6, 508 passim. doi: 10.1016/s0001-2092(07)66673-3. No abstract available. PMID 2467620